CLINICAL TRIAL: NCT03970629
Title: ROSA Total Knee Investigational Testing Authorization Study: Prospective Single Center Study of the ROSA Total Knee System
Brief Title: ROSA Total Knee Investigational Testing Authorization Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenging enrollment due to COVID-19.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEU2018-46K
Record Dates: First submitted 2019-05-30; First posted 2019-05-31 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Knee Pain; Chronic Osteoarthritis; Avascular Necrosis of Femoral Condyle; Moderate Varus, Valgus or Flexion Deformities; Rheumatoid Arthritis
MeSH Terms: conditions — Genu Valgum; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Assisted TKA (Active Comparator): Robotic Assisted TKA via ROSA Robot
  Interventions: Device: PERSONA Total Knee
- Conventional TKA (Active Comparator): Conventional TKA
  Interventions: Device: PERSONA Total Knee

INTERVENTIONS:
Device: PERSONA Total Knee — Primary Total Knee Arthroplasty

SUMMARY:
This is a prospective, single-center clinical study designed to facilitate the collection and evaluation of workflow efficiency, patient pain and function, and adverse event data. This clinical study will include Persona Total Knee components using the ROSA Total Knee Robotic System or conventional instrumentation.

DETAILED DESCRIPTION:
The primary objective of this study is to collect and compare clinical outcomes and surgical data using the ROSA Total Knee robotic instrumentation and conventional instrumentation in primary total knee arthroplasty.

The assessments will include: Planned vs actual component positioning; Workflow efficiency; Patient safety based on incidence and frequency of adverse events; Clinical performance measured by overall pain and function, quality of life data, and radiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is a minimum of 18 years of age
2. Pre-op component positioning and sizing plan prior to surgery
3. Independent of study participation, patient is a candidate for primary TKA using the commercially available Persona knee components implanted in accordance with product labeling
4. Patient has participated in this study-related Informed Consent process
5. Patient is willing and able to provide written Informed Consent by signing and dating the IRB or EC approved Informed Consent form
6. Patient is willing and able to complete scheduled study procedures and follow-up evaluations

Exclusion Criteria:

1. Patient is currently participating in any other surgical intervention studies or pain management studies
2. Patient has underwent contralateral UKA or TKA within the last 18 months
3. Hip pathology with significant bone loss (e.g. avascular necrosis of the femoral head with collapse, severe dysplasia of the femoral head or the acetabulum)
4. Hip pathology severely limiting range of motion (e.g. arthrodesis, severe contracture, chronic severe dislocation)
5. Patient is pregnant or considered a member of a protected population (e.g., prisoner, mentally incompetent, etc.)
6. Patient has previously received partial or total knee arthroplasty for the ipsilateral knee

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
EQ-5D questionnaire | 1 year
  EQ-5D
Oxford Knee Score Questionnaire | 1 year
  Oxford Knee Score

CONTACTS AND LOCATIONS:
Overall Officials: Charles Jaggard, Study Director — Zimmer Biomet
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No